CLINICAL TRIAL: NCT02407821
Title: A Pilot Study to Evaluate the Feasibility and Safety of Performing a Double Blind, Placebo-controlled, Randomized Controlled Trial of the Routine Use of SSRI's at the Initiation of End-stage Renal Disease Treatment
Brief Title: The Routine Use of SSRI's at the Initiation of End-stage Renal Disease Treatment (RoSIE)
Acronym: RoSIE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor enrolment
Sponsor: University Health Network, Toronto (Other)
Collaborators: McMaster University (Other); Unity Health Toronto (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2015-03-16; First posted 2015-04-03 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-09

CONDITIONS: End Stage Renal Disease
Keywords: Controlled Clinical Trials, Randomized; Kidney Failure; Renal Insufficiency, Chronic; Dialysis, Renal; Peritoneal Dialysis; Hemodialysis; Depressive Symptoms; Selective Serotonin Reuptake Inhibitors; Antidepressants; Escitalopram
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency; Renal Insufficiency, Chronic; Depression | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Escitalopram (Active Comparator)
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram — Dose will be initiated at 5 mg daily. At two weeks, a safety and tolerability assessment will be performed, and if tolerated, the dose will be increased to 10 mg daily. At 24 weeks, the medication will be titrated downwards to 5 mg daily for a further two weeks before discontinuation.
  Arms: Escitalopram
Drug: Placebo — The matching placebo will be up-titrated and down-titrated at the same time intervals as the active medication.
  Arms: Placebo

SUMMARY:
In this study the investigators hypothesize that antidepressant therapy may improve the overall welling of patients with acute or chronic kidney disease when given around the time of starting chronic dialysis therapy. This study is a pilot, randomized controlled trial that aims to examine whether prescribing oral escitalopram to all incident dialysis patients is safe and feasible.

DETAILED DESCRIPTION:
Over 120,000 people with kidney disease start chronic dialysis therapy across North America each year. In addition to high mortality, studies uniformly report high rates of depression, pain and non-specific symptoms after dialysis is started. Suicide rates are high, particularly early in the treatment history, and withdrawal from dialysis is increasingly common in recent years, suggesting a high burden of depressive symptoms. While various treatments appear to be effective, there are multiple barriers preventing patients from getting or accepting appropriate care for depression. The investigators hypothesize that antidepressant therapy may improve morbidity and mortality when prescribed to patients with acute or chronic kidney disease (CKD) around the time of starting chronic dialysis therapy.

This is a phase II, multi-centre, double blind, randomized controlled trial to compare the safety and feasibility of oral escitalopram to placebo in incident dialysis patients. Those who have started chronic dialysis therapy within 12 weeks of being identified will be eligible for the study. Participants will randomized 1:1 to receive either escitalopram or placebo daily for 26 weeks.

The primary outcome is feasibility in terms of recruitment rates and protocol compliance. The secondary outcomes include estimates of safety (adverse events) and efficacy (hospitalization days, mortality, and changes in depression and quality of life scores). This pilot trial is intended to guide and inform the design of a full scale study to evaluate whether the routine use of escitalopram can improve the quality of life and hospital free days in patients on dialysis, as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female aged ≥ 25 years
2. Patient or substitute decision maker willing and able to give informed consent
3. Incident to dialysis defined as within a 12-week window from the first dialysis treatment (1 week prior to, to 11 weeks after). Patients on all forms of dialysis except CRRT (including peritoneal dialysis, home hemodialysis, in-centre intermittent hemodialysis and nocturnal dialysis) will be eligible. Patients returning to dialysis after transplant graft loss will be eligible.

Exclusion Criteria:

1. Past history of allergy to, or intolerance of, escitalopram
2. Known severe hepatic dysfunction
3. Recent history of active bleeding within the past 3 months (e.g. gastrointestinal bleeding requiring hospitalization) or known bleeding disorder
4. Current use of class I anti-arrhythmic medications; SSRI or SNRI antidepressants; pimozide, MAO inhibitors, reserpine, guanethidine, cimetidine or methyldopa, omeprazole; tri-cyclic and tetra-cyclic anti-depressants, neuroleptics or anti-convulsants, triptans, tramadol, linezolid, tryptophan, and St. John's Wort; but not gabapentin
5. Past treatment failure for depression with escitalopram or with ≥ 2 antidepressant treatments of at least 6 weeks duration each
6. Initiation of psychotherapy for depression in the 3 months prior to study entry
7. Alcohol or substance abuse or dependence that requires acute detoxification at study entry
8. Present or past psychosis or bipolar disorder, schizophrenia or any other psychotic disorder documented in medical records
9. Suicidal ideation defined as the patient is at significant risk of suicide on the Columbia Suicide Scale71 or has attempted suicide within 6 months prior to the Screening Visit
10. Clinically-identified major depressive disorder that, in the opinion of the clinical team, requires treatment
11. Pregnancy, lactation and women of childbearing potential not using adequate contraception
12. Abnormal QTc at baseline: QTcF interval >600 ms (based on the Fredericia correction where QTcF = QT/RR0.33)66
13. Lactose intolerance (as placebo contains lactose)
14. Known uncontrolled glaucoma
15. Patients requiring treatment with continuous renal replacement therapy (CRRT)
16. Documented history of brain tumour

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Proportion of consecutive incident dialysis patients that are eligible | 12 months
Proportion of eligible patients that will consent to randomization | 12 months
Proportion of randomized patients that comply with their group assignment | 12 months
  Compliance defined as >80% of doses taken

SECONDARY OUTCOMES:
Serious adverse events | 12 months
Number of patients withdrawn from the study drug due to QTc prolongation | 12 months
Completion rate for all secondary outcome measures (KDQoL, HUI-III, PHQ-9, Handgrip and 2-Minute Walk Test) | 3 months and 6 months
Death | 12 months
Hospital-free days | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Vanita Jassal, MD, Principal Investigator — University Health Network, Toronto
Locations (3):
- Canada (3):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario